CLINICAL TRIAL: NCT02656784
Title: The Resonance Assessment in Magnetic Measurement of the Effect of Psychotherapy in Obsessive-compulsive Disorder in a Randomized Clinical Trial
Brief Title: The Efficacy of TBCT Compared to ERP in the Treatment of OCD Patients, by the Assessment of Magnetic Resonance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do PiauÍ (Other)
Collaborators: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Eleonardo Pereira Rodrigues, Effective Professor of Psychology Course. Coordinator of the Cognitive Neuroscience Laboratory., Universidade Estadual do PiauÍ
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UESPI
Record Dates: First submitted 2015-12-05; First posted 2016-01-15 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: OBSESSIVE COMPULSIVE DISORDER (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Behavior Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Trial-Based Cognitive Therapy (TBCT) (Experimental): Trial-Based Cognitive Therapy (TBCT) is a three-level, three-phase, case formulation approach, based on the work of Franz Kafka "The Trial" and developed by Professor Irismar Reis de Oliveira at Federal University of Bahia, Brazil. TBCT's foundation is in cognitive therapy (CT); however, it has a unique approach to conceptualization and techniques that make it a distinct intervention in modifying patients' core beliefs, especially those about the self. All individuals in the group will be submitted to MRI
  Interventions: Behavioral: Behavioral Therapy
- Behavioral Therapy (ERP) (Experimental): The Behavioral Therapy is an intervention of first choice for treatment of OCD , which employs the technique of Exposure and Response Prevention (ERP) , considered the gold standard to the disorder. The technique involves directly exposing patients to recall stimulation of obsessive thoughts and prevent them from performing the compulsive rituals. All individuals in the group will be submitted to MRI
  Interventions: Behavioral: Cognitive Therapy
- Control Group (No Intervention): The control group consisted of individuals without OCD, matched with the experimental group in terms of gender,age and education. In this group are not included in individuals in psychotherapeutic care and with a history of neurological or psychiatric disorder; however, all them will be submitted to MRI .

INTERVENTIONS:
Behavioral: Cognitive Therapy — Trial-Based Cognitive Therapy (TBCT) is a three-level, three-phase, case formulation approach. TBCT's foundation is in cognitive therapy (CT); however, it has a unique approach to conceptualization and techniques that make it a distinct intervention in modifying patients' core beliefs, especially those about the self. All the individuals will be submitted to MRI.
  Other Names: Trial-based cognitive therapy
  Arms: Behavioral Therapy (ERP)
Behavioral: Behavioral Therapy — The Behavioral therapy employs the technique of Exposure and Response Prevention ( ERP ).The technique involves directly exposing patients to recall stimulation of obsessive thoughts and prevent them from performing the compulsive rituals. All the individuals will be submitted to MRI.
  Other Names: Exposure and Response Prevention (ERP)
  Arms: Trial-Based Cognitive Therapy (TBCT)

SUMMARY:
This is a sample made up of ninety-six adult individuals of both sexes to be divided into three groups: the experimental group of thirty-two patients with OCD who will be undergone Trial-Based Cognitive Therapy; the gold standard, with thirty-two people with OCD subject Exposure and Response Prevention and the control group of thirty-two healthy individuals. Interviews and therapeutic intervention occur in private practices researchers or medical schools accredited by UESPI.

Experimental group: Will be eligible adults of both sexes with educational level equal to or higher education complete primary, aged between 18 and 60 years with OCD diagnosis confirmed according to criteria DSM-IV (APA, 1994). It is going to be excluded patients who had previously undergone treatment behavioral psychotherapy or cognitive-behavioral approach.

DETAILED DESCRIPTION:
OBJECTIVES

Evaluate the effectiveness of Trial-Based Cognitive Therapy (TBCT) compared to Exposure and Response Prevention (ERP) in the treatment of OCD patients, by neuroimaging tests such as MRI.

1. Describe the neuroanatomical profile of the sample participants before and after the psychotherapeutic intervention by MRI;
2. Compare the profile neuroanatomical between the experimental group and the control group by MRI;
3. Identify possible neuroanatomical differences in the participating sample of pre and post-treatment, both among individuals and among psychotherapeutic intervention groups;
4. To investigate associations between the results of MRI scans and indexes the scales currently used to assess severity of OCD.

ELIGIBILITY:
Inclusion Criteria:

* Will be eligible adults of both sexes with educational level equal to or higher education complete primary, aged between 18 and 60 years with OCD diagnosis confirmed according to criteria DSM-IV

Exclusion Criteria:

* It is going to be excluded patients who had previously undergone treatment behavioral psychotherapy or cognitive-behavioral approach.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
The severity of OCD (Morphological and physiological changes in the brain) | 12 weeks (3 months)
  Data colected at 1st week, 6th week, 12th week. Scales used are Yale-Brown Obssessive Compulsive Scale and Symptoms of Checklist (Y-BOCS), Beck Depression Inventory (BDI), Beck Anxienty Inventory (BAI), Obsessive-Compulsive Beliefs Questionnaire-87 (OBQ-87), The Medical Outcomes Study 36 - Item Short Form Health Survery ( SF-36), Questionnare of Cognitive Distortions (CD-Quest), Subjective Units of Discomfort (SUDS) and MRI.

SECONDARY OUTCOMES:
Quality of Life | 12 weeks
  Data colected at 1st week and 12th week and, at follow-up, after three months, six months and one year. The scale used is SF-36
Quality of Life | 1 year
  At follow-up, after three months, six months and one year. The scale used is SF-36
Cognitive Distortions | 12 weeks
  Data colected every week (during 12 weeks). The scale used is CD-Quest
Cognitive Distortions | 1 year
  At follow-up, after three months, six months and one year. The scale used is Cognitive Distortions Questionnaire.
Severity of OCD | 12 weeks
  Data colected at 1st week, 6th week and 12th week and, at follow-up, after three months, six months and one year. The scale used is Y-BOCS
Severity of OCD | 1 year
  At follow-up, after three months, six months and one year. The scale used is Y-BOCS.
The Assessment of Depression | 12 weeks
  Data colected at 1st week, 6th week and 12th week and, at follow-up, after three months, six months and one year. The scale used is BDI
The Assessment of Depression | 1 year
  At follow-up, after three months, six months and one year. The scale used is BDI
The Assessment of Anxiety | 12 weeks
  Data colected at 1st week, 6th week and 12th week and, at follow-up, after three months, six months and one year. The scale used is BAI
The Assessment of Anxiety | 1 year
  At follow-up, after three months, six months and one year. The scale used is BAI
The Assessment of Magnetic Resonance (MRI) | 15 weeks
  Data colected at zero week and 15th week. The scale used is MRI
The Assessment of The Obssessive Beliefs | 15 weeks
  Data colected at zero week and 15th week. The scale used is OBQ-87
The level of Anxiety (Obssessive, Compulsive and Evitation Symptoms) | 12 weeks
  Data colected every week (during 12 weeks). The scale used is SUDS

CONTACTS AND LOCATIONS:
Overall Officials: Eleonardo P Rodrigues, Psy MSc, Principal Investigator — Piaui State University - Brazil - UESPI - Recruiting; Irismar R De Oliveira, PhD, Study Director — Bahia Federal University - Brazil - UFBA
Locations (1):
- Piauí State University - UESPI, Teresina, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No